CLINICAL TRIAL: NCT00909116
Title: International Transtar Registry - Stapled Transanal Rectal Resection Performed With Contour Transtar Stapler in the Treatment of Obstructed Defecation Syndrome (ODS)
Brief Title: International Multicenter Prospective Transtar Registry
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Europe) GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CME-08-001
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Constipation
Keywords: ODS; chronic constipation; internal rectal prolapse; rectocele; Stapled Transanal Rectal Resection; Contour Transtar; STARR
MeSH Terms: conditions — Constipation; Rectocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Chronic constipation - ODS: Adult Patients with ODS
  Interventions: Procedure: Stapled Transanal Rectal Resection with Contour Transtar

INTERVENTIONS:
Procedure: Stapled Transanal Rectal Resection with Contour Transtar — Transanal Stapling procedure - Stapled Transanal Rectal Resection

SUMMARY:
Obstructed Defecation Syndrome (ODS) describes a condition which is characterized by chronic constipation. The symptoms of ODS include abdominal pain or cramping, irregular bowel frequency and the feeling of not having emptied the rectum. ODS is usually associated with internal rectal prolapse and/or rectocele. For surgical treatment of ODS, a plethora of surgical techniques have been described with no one method having been assessed as a gold standard.

DETAILED DESCRIPTION:
A new surgical procedure - Transtar - has been introduced in Europe recently. The goal of this registry is to assess safety, effectiveness and patient quality of life, associated with Transtar for chronic constipation due to morphological changes, such as internal rectal prolapse and rectocele.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obstructed defecation, fragmented defecation or incomplete evacuation as a presenting symptom documented by a standardized symptom score
* confirmed internal rectal prolapse or rectocele on dynamic defecography
* adequate external sphincter on rectal digital examination.

Exclusion Criteria:

* Subjects with any other surgical procedure than STARR for ODS
* Subjects in whom STARR is not performed with the Contour Transtar stapler
* Subjects with a physical or psychological condition which would impair participation in the registry.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive male and female patients of at least 16 years with symptoms of chronic constipation due to ODS associated with anatomical changes, such as internal rectal prolapse and rectocele
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-01-31 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Change in constipation symptoms measured by KESS score | preoperative, and at 12 months post-op

SECONDARY OUTCOMES:
Changes in patients symptoms measured by Incontinence score and ODS Score, QoL measures with EQ5D and PAC-QoL | preoperative, at 6 weeks and 12 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Goran Ribaric, MD,PhD, Study Director — Ethicon Endo-Surgery (Europe) GmbH
Locations (1):
- Andree D'Hoore, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
via publication

REFERENCES:
- [Background] Schwandner O, Stuto A, Jayne D, Lenisa L, Pigot F, Tuech JJ, Scherer R, Nugent K, Corbisier F, Basany EE, Hetzer FH. Decision-making algorithm for the STARR procedure in obstructed defecation syndrome: position statement of the group of STARR Pioneers. Surg Innov. 2008 Jun;15(2):105-9. doi: 10.1177/1553350608316684. Epub 2008 Apr 9. PMID 18403378
- [Background] Renzi A, Talento P, Giardiello C, Angelone G, Izzo D, Di Sarno G. Stapled trans-anal rectal resection (STARR) by a new dedicated device for the surgical treatment of obstructed defaecation syndrome caused by rectal intussusception and rectocele: early results of a multicenter prospective study. Int J Colorectal Dis. 2008 Oct;23(10):999-1005. doi: 10.1007/s00384-008-0522-0. Epub 2008 Jul 25. PMID 18654789